CLINICAL TRIAL: NCT05830669
Title: Effect of Remote Ischemic Preconditioning in Septic Patients on Cell Cycle Arrest Biomarkers - the RIPC-ICU Randomized Clinical Trial
Brief Title: Remote Ischemic Preconditioning in Septic Patients
Acronym: RIPC-ICU
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universität Münster (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: AnIt22-06
Record Dates: First submitted 2023-03-30; First posted 2023-04-26 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Critically Ill; Acute Kidney Injury; Sepsis
MeSH Terms: conditions — Critical Illness; Acute Kidney Injury; Sepsis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Remote ischemic preconditioning (RIPC) Three Cycles of 5-min upper limb ischemia. If there is no response this will be followed by 2 cycles of 10-min upper-limb ischemia.
  Interventions: Procedure: Remote ischemic preconditioning (RIPC)
- Control Group (Sham Comparator): Three cycles of 5- min upper limb sham ischemia.
  Interventions: Procedure: Sham RIPC

INTERVENTIONS:
Procedure: Remote ischemic preconditioning (RIPC) — 3 cycles of 5 min inflation of a blood-pressure cuff to 200 millimetres of mercury (mmHG) (or at least to a pressure 50 mmHG higher than the systolic arterial pressure) to one upper arm followed by 5 min reperfusion with the cuff deflated. In Non-Responder two additional cycles of 10 min cuff inflation will be performed.
  Arms: Intervention Group
Procedure: Sham RIPC — 3 cycles of 5 min inflation of a blood-pressure cuff to 20 mmHG to one upper arm followed by 5 min reperfusion with the cuff deflated. In Non-Responder two additional cycles of 10 min cuff inflation will be performed
  Arms: Control Group

SUMMARY:
Acute kidney injury is a well-recognized complication in critically ill patients. Up to date there is no clinically established method to reduce the incidence or the severity of acute kidney injury.

Remote ischemic preconditioning (RIPC) will be induced by three cycles of upper limb ischemia.

The aim of the study is to reduce the incidence of AKI by implementing remote ischemic preconditioning (identified by the urinary biomarkers tissue inhibitor of metalloproteinases-2 (TIMP-2) and insulin-like growth factor-binding protein 7(IGFBP7)

DETAILED DESCRIPTION:
Acute kidney injury (AKI) is a common complication in critically ill patients with sepsis. To date, there is no pharmacological option to treat or prevent AKI.

Ischemic conditioning is an innate tissue adaptation elicited by ischemia that mediates local and remote organ protection against subsequent exposure to the same or other injury.

The aim of this trial is to evaluate the effects of remote ischemic conditioning in critically ill patients on acute kidney injury.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age ≥18 years)
* Critically ill patients with sepsis < 12 hours
* Invasive ventilation for at least 24 hours (propofol-free-sedation) and/or vasopressor therapy
* Unrestricted intensive care for at least 72 hours
* Written informed consent

Exclusion Criteria:

* Pre-existing AKI
* (Glomerulo-)nephritis, interstitial nephritis, vasculitis
* Chronic kidney disease with estimated glomerular filtration rate (eGFR) < 30 ml/min/1.73m²
* Chronic dialysis dependency
* Kidney transplant in the last 12 months
* Oral antidiabetics, sulfonamides or nicorandil
* Pregnancy or breastfeeding
* Do-not-reanimate order
* Participation in another interventional trial involving kidney outcomes within the last 3 months
* Dependency on the investigator or center

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2023-05-11 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
1. kidney damage after cardiac surgery identified by the difference between [TIMP-2]*[IGFBP7] levels 24h after randomization and [TIMP-2]*[IGFBP7] levels at randomization | from randomization to 24 hours after randomization

SECONDARY OUTCOMES:
Incidence of Acute Kidney Injury (AKI) according to the Kidney Disease: Improving Global Outcomes (KDIGO) criteria | 72 hours after the onset of sepsis
Severity of AKI | 72 hours after the onset of sepsis
  The severity for AKI is classified according to the KDIGO criteria
Need for renal replacement therapy | 72 hours after the onset of sepsis
  Number of patients with renal replacement therapy
Recovery of kidney function | day 90 after the onset of sepsis
  defined as complete recovery: serum-creatinine ≤0.5 mg/dl higher than baseline; partial recovery: serum creatinine >0.5 mg/dl higher than baseline but no dialysis-dependence; non-recovery: patients who remained dialysis-dependent
Mortality | day 90 after the onset of sepsis
Major adverse kidney events (MAKE) Composite endpoint consisting of death, renal replacement therapy, and persistent severe AKI lasting for 72 hours or more | day 90 after the onset of sepsis
Length of Intensive Care Unit (ICU) stay | up to 90 days after onset of sepsis
Length of hospital stay | up to 90 days after onset of sepsis

OTHER OUTCOMES:
Add-on Study (Analysis of further proteins) | from randomization until 24 hours after randomization

CONTACTS AND LOCATIONS:
Overall Officials: Melanie Meersch-Dini, MD, Principal Investigator — University Hospital Muenster, Dept. of Anesthesiology, Intensive Care Therapy and Pain Medicine
Locations (1):
- University Hospital Münster; Department of Anesthesiology, Intensive Care Medicine and Pain Medicine, Münster, Germany

IPD SHARING:
Plan to Share IPD: No